CLINICAL TRIAL: NCT01563198
Title: Amelioration of Claustrophobia and Disruptive Patient Motion in MR Imaging
Brief Title: Reduction of Claustrophobia and Patient Motion After Training of MRI Personnel in Comfort TalkTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hypnalgesics, LLC (Industry)
Collaborators: Tufts Medical Center (Other); Boston Medical Center (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R43AT0062696
Record Dates: First submitted 2011-10-24; First posted 2012-03-26 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Claustrophobia; Complication of Diagnostic Procedure
Keywords: MRI departments and facilities; Noncompletion of MRI
MeSH Terms: conditions — Claustrophobia | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Comfort Talk® Training (Experimental): The MRI units of three clinical sites form the group. Their personnel will be trained to use Comfort Talk® to help patients who are claustrophobic, anxious, and/or cannot lie still to complete their tests
  Interventions: Behavioral: Comfort Talk®

INTERVENTIONS:
Behavioral: Comfort Talk® — Personnel of MRI units will be trained in advanced rapport skills, patient-centered and hypnoidal language, correct use of suggestions and skills of tension diffusion. This will entail 16 hrs class room work, additional on-site post-training support, and access to a post-training support web module resulting in at least 20 hrs training.
  Other Names: Self-hypnotic relaxation; nonpharmacologic analgesia; nonpharmacologic anxiolysis; patient sedation without medication

SUMMARY:
Annually, an estimated 700,000 patients do not complete their scheduled MRI scans because of claustrophobia or inability to hold still. Training staff working in MRI facilities to provide Comfort Talk® promises to enable patients to complete and obtain high quality imaging without medication, which will increase comfort and reduce sedation risks for the patients, and increase efficiency and reduce loss of revenue for the facilities.

DETAILED DESCRIPTION:
Claustrophobia and disruptive patient motion are common impediments to MRI examination, but they may be prevented or ameliorated with a non-pharmacologic behavioral intervention administered by trained staff. The potential benefits of such an intervention are highly significant, considering that the alternatives are to cancel the study or administer sedation. Inability to complete their MRI scans adversely affects an estimated 700,000 patients every year in the US. These patients are either deprived of a diagnosis, subject to diagnostic delays, or are exposed to risks of pharmacologic sedation, including death. The imaging facilities in turn, typically cannot fill the suddenly vacated examination slots in time before the next scheduled patient and thus incur considerable lost revenue and efficiency. The long-term goal is to provide a validated, clinically feasible means for non-pharmacologic amelioration of claustrophobia and disruptive patient motion, achieved by training MRI staff to use advanced rapport skills and comforting language to help patients. Phase I will design and perform a formative evaluation of a Comfort Talk® Training intervention so that definitive testing of the hypothesized benefits for the intervention can be accomplished in Phase II.

In Specific Aim 1 the Comfort TalkTM intervention sequence will be designed to include training in advanced rapport skills, using basic comforting language and avoiding negative language for all facility staff (including receptionists, technologists, nurses, and physicians). A core of licensed healthcare professionals will be taught how to guide patients in self-hypnotic relaxation techniques, using scripts, found to be safe and effective in the radiology department. Techniques are designed to easily integrate into the normal workflow without adding time. Training will include 2x8 hrs live at three test sites. Acceptance, observation of staff behavior, qualitative feedback, and rates of noncompletion will be used to assess efficacy of training, guide prototype development, and develop train-the-trainer materials. Using in-market piloting techniques, niche applications with their metrics will be explored to develop situation-specific supplemental materials. In Aim 2 an interactive web-based electronic platform will be developed to supplement training and provide post-training support. It will provide scenarios and practice applications, guided dialogue options, functions for online live interactive classes, and interface with smartphones. The prototype will be beta-tested with 20 experts in hypnosis and refined through user input from the test sites. Aim 3 is to conduct a formative evaluation of the entire Comfort Talk® intervention. Effects will be evaluated in 3-months intervals and compared to baseline performance. Criteria will include acceptance, qualitative feedback, content mastery, staff behavior, rates of noncompletion, patient recall and satisfaction. Additional metrics identified through in-market exploration will be analyzed for their potential as economic drivers and evaluation instruments.

ELIGIBILITY:
Inclusion Criteria:

* Facilities performing MRI examinations
* Facilities capturing data on noncompletion of MRI scans
* Facilities willing to have their personnel trained
* Facilities with personnel interested and willing to be trained
* Facilities able to obtain IRB review

Exclusion Criteria:

* Facilities not performing MRI examinations
* Facilities not capturing data on noncompletion of MRI scans
* Facilities not willing to have their personnel trained
* Facilities unable to obtain IRB review

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97712 (Actual)
Dates: Start 2011-08; Primary Completion 2015-07 (Actual); Study Completion 2016-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira V Lang, MD, Principal Investigator — Hypnalgesics, LLC
Locations (4):
- United States (4):
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Hypnalgesics, LLC, Brookline, Massachusetts
  - Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang EV, Ward C, Laser E. Effect of team training on patients' ability to complete MRI examinations. Acad Radiol. 2010 Jan;17(1):18-23. doi: 10.1016/j.acra.2009.07.002. Epub 2009 Sep 5. PMID 19734060
- [Background] Lang EV, Benotsch EG, Fick LJ, Lutgendorf S, Berbaum ML, Berbaum KS, Logan H, Spiegel D. Adjunctive non-pharmacological analgesia for invasive medical procedures: a randomised trial. Lancet. 2000 Apr 29;355(9214):1486-90. doi: 10.1016/S0140-6736(00)02162-0. PMID 10801169
- [Result] Norbash A, Yucel K, Yuh W, Doros G, Ajam A, Lang E, Pauker S, Mayr N. Effect of team training on improving MRI study completion rates and no-show rates. J Magn Reson Imaging. 2016 Oct;44(4):1040-7. doi: 10.1002/jmri.25219. Epub 2016 Apr 6. PMID 27126735
- [Result] Lang EV, Yuh WT, Ajam A, Kelly R, Macadam L, Potts R, Mayr NA. Understanding patient satisfaction ratings for radiology services. AJR Am J Roentgenol. 2013 Dec;201(6):1190-5; quiz 1196. doi: 10.2214/AJR.13.11281. PMID 24261356
- See also: Explanation of Comfort TalkTM and access to Post-Training Support Module — http://www.ComfortTalk.com
- See also: Sponsor website and background information; description of techniques used — http://ComfortTalk.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Different participants were assessed at baseline and after training.
Units Other Than Participants: Clinical sites
Groups:
- Comfort TalkTM Training: The MRI units of three clinical sites form the group. Their personnel will be trained to use Comfort TalkTm to help patients who are claustrophobic, anxious, and/or cannot lie still to complete their tests
  Comfort Talk: Personnel of MRI units will be trained in advanced rapport skills, patient-centered and hypnoidal language, correct use of suggestions and skills of tension diffusion. This will entail 16 hrs class room work, additional on-site post-training support, and access to a post-training support web module resulting in at least 20 hrs training.
Period: Baseline
Arm/Group | Comfort TalkTM Training
Started | 49733; 3 Clinical sites
Completed | 49733; 3 Clinical sites
Not Completed | 0; 0 Clinical sites
Period: After Training
Arm/Group | Comfort TalkTM Training
Started | 47979; 3 Clinical sites
Completed | 47979; 3 Clinical sites
Not Completed | 0; 0 Clinical sites

BASELINE CHARACTERISTICS:
Population: We obtained cumulative data from patients completion rates, thus no individual patient data on age, gender, ethnicity are available. MR departments per se do not have personal characteristics.
Units Other Than Participants: MRI sites
Groups:
- Comfort Talk® Training: The MRI units of three clinical sites form the group. Their personnel will be trained to use Comfort TalkTm to help patients who are claustrophobic, anxious, and/or cannot lie still to complete their tests
  Comfort Talk: Personnel of MRI units will be trained in advanced rapport skills, patient-centered and hypnoidal language, correct use of suggestions and skills of tension diffusion. This will entail 16 hrs class room work, additional on-site post-training support, and access to a post-training support web module resulting in at least 20 hrs training.
Arm/Group | Comfort Talk® Training
Number analyzed (Participants) | 49733
Number analyzed (MRI sites) | 3
Age, Categorical [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: We obtained cumulative data from patients' show-up and completion rates, thus no individual patient data on age, gender, ethnicity are available. MR departments per se do not have personal characteristics.
  Participants
    number analyzed (Participants) | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: We obtained cumulative data from patients' show-up and completion rates, thus no individual patient data on age, gender, ethnicity are available. MR departments per se do not have personal characteristics.
  Participants
    number analyzed (Participants) | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
No-show rate [Number; unit: Percentage of participants] | 11.2
Non-completion rate of showing-up patients [Number; unit: Percentage of all showing-up patients] — Population: Participants were from 3 MRI sites whose teams were trained in Comfort Talk®. In this analysis only patients who showed up at the MRI sites at baseline were included (all participants - no-shows).
  Percentage of all showing-up patients
    number analyzed (Participants) | 44140
    (all) | 2.3
Non-completion rate of all scheduled patients [Number; unit: Percentage of all scheduled participants] — Participants were from 3 MRI sites whose teams were trained in Comfort Talk®. In this analysis all patients scheduled for an MRI at baseline were included as denominator.
  Percentage of all scheduled participants | 13.3

OUTCOME MEASURES:

1. Primary Outcome: Change in Non-completion Rate of MRI Scans From the Average of the Baseline Year to the Average of One Year Post Training (All Scheduled Patients)
Description: The sites will be followed for an average of one year after training in Comfort Talk and non-completion rates will be compared to the baseline values of non-completion among all scheduled patients.
Time Frame: Baseline average of one year plus post training average one year = 2 years
Population: Participants were from MRI 3 sites whose teams were trained in Comfort Talk®. In this analysis all patients who were scheduled for scans during the baseline year and the year after training were included
Measure: Number; unit: Percentage of participants
Arm/Group | Comfort TalkTM Training
Number analyzed (Participants) | 97712
Percentage of participants
  Non-completion Rate after Training: number analyzed (Participants) | 47979
  Non-completion Rate after Training | 10
  Change from Baseline | -3.3
Statistical Analysis 1: Comparison: Comfort TalkTM Training; Change in Non-completion Rate of MRI Scans From Baseline at Average of One Year (All Schedule Patients); Test type: Superiority; p < 0.0001, Chi-squared

2. Primary Outcome: Change in Non-completion Rate of MRI Scans From the Average of the Baseline Year to the Average of One Year Post Training (Showing-Up Patients Only)
Description: The change in non-completion rate of MRI scans, obtained for the year prior to Comfort Talk® training at baseline, to the average one year post training was assessed
Time Frame: Baseline average of one year plus post training average one year = 2 years
Population: Participants were from 3 MRI sites whose teams were trained in Comfort Talk®. In this analysis only patients who showed up at the MRI sites at baseline year and the year after training were included (all participants minus no-shows).
Measure: Number; unit: Percentage of showing-up participants
Arm/Group | Comfort TalkTM Training
Number analyzed (Participants) | 87956
Percentage of showing-up participants
  Non-Completion Rate after Training: number analyzed (Participants) | 43816
  Non-Completion Rate after Training | 1.4
  Change from Baseline | -0.9
Statistical Analysis 1: Comparison: Comfort TalkTM Training; Test type: Superiority; p < 0.0001, Chi-squared

3. Secondary Outcome: Change in No-Show Rates of Patients From the Average of the Baseline Year to the Average of One Year Post Training
Description: The sites will be followed for an average of one year after training in Comfort Talk and no-show rates will be compared to the baseline values of non-completion among all scheduled patients which were also collected over 1 year.
Time Frame: Baseline average of one year plus post training average one year = 2 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Comfort TalkTM Training
Number analyzed (Participants) | 97712
Percentage of participants
  No-Show Rate After Training: number analyzed (Participants) | 47979
  No-Show Rate After Training | 8.7
  Change From Baseline | -2.5
Statistical Analysis 1: Comparison: Comfort TalkTM Training; Test type: Superiority; p < 0.0001, Chi-squared

ADVERSE EVENTS:
Time Frame: One year starting with the training
Description: Adverse events were monitored during the training days of the MRI teams. Then assessment was non-systematic in that we would have reported adverse events if they had become known or being collected after training. Patients at risk were only those in the post-training period who showed up at the facility including those who completed their scans and also those who did not.
Arm/Group | Comfort TalkTM Training
Serious Adverse Events (participants affected / at risk) | 0/43816
Other Adverse Events (participants affected / at risk) | 0/43816

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No